CLINICAL TRIAL: NCT05773157
Title: Evaluation of SNAP-Ed Online Modules to Improve Responsive Feeding Practices of Caregivers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Jennifer Savage Williams, Director Center For Childhood Obesity Research, Penn State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00020516
Record Dates: First submitted 2023-03-06; First posted 2023-03-17 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Feeding Behavior
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: A single pilot group of participants will complete the online modules and evaluate their effectiveness using pre and post surveys.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Receive Online Modules (Other): All participants receiving the same online modules intervention.
  Interventions: Behavioral: Online Modules

INTERVENTIONS:
Behavioral: Online Modules — Participants receive modules to improve responsive feeding practices of caregivers

SUMMARY:
Evaluation of three online modules developed by the Center for Childhood Obesity Research for caregivers of children ages 5-12 years old participating in SNAP-Ed programing.

DETAILED DESCRIPTION:
the Center for Childhood Obesity Research developed three online modules for caregivers of children ages 5-12 years old who are participating in SNAP-Ed programming. These modules were developed to be used within the context of normal programming that participants will receive in any given year. The specific aim are as follows:

Aim #1: To examine acceptability of these modules by caregivers participating in SNAP-Ed programming. This will be assessed by evaluating acceptability questions answered by participants after completing the modules.

Aim #2: To examine the feasibility of these modules by caregivers participating in SNAP-Ed programming, assessed by >60% completion rate of all three modules.

Online module content will focus on topics such as:

* Shared Responsibility of Feeding:
* Parent Provides, Child Decides
* Family Mealtimes
* Hunger and Fullness
* Avoiding use of controlling feeding practices

ELIGIBILITY:
Inclusion Criteria:

* Primary caregiver of a child between the ages of 2 to 16 years
* Over the age of 18
* English-speaking
* Have a reliable internet source and active email account so they can access the online modules

Exclusion Criteria:

* Are not the primary caregivers of a child between the ages of 2 to 16 years
* Are under the age of 18
* Are not English-speaking
* Do not have a reliable internet source or email address

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Feeding Practices | 1 month
  Pre/post Feeding Practices surveys

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared